CLINICAL TRIAL: NCT05960812
Title: Skillful Neglect Vs Repair For Upper Border Subscapularis Tear Associated With Posterosuperior Cuff Tears Repair In Non-Athletes: A Randomized Controlled Trial
Brief Title: Skillful Neglect Vs Repair For Subscapularis Tear Associated With Posterosuperior Cuff Tears Repair.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohamed Ashraf Abdallah (Other)
Responsible Party: Sponsor-Investigator, Mohamed Ashraf Abdallah, Principal investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MD 218/2022
Record Dates: First submitted 2023-05-20; First posted 2023-07-27 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Subscapularis Muscle Strain
Keywords: Rotator cuff tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (patient treated by skillful neglect with biceps tenotomy) (Active Comparator): neglect of upper border subscapularis tear and doing biceps tenotomy
  Interventions: Procedure: skillful neglect Of upper subscapularis tear in Lafosse type 1 and type 2 with long head biceps tenotomy .; Procedure: arthroscopic repair Of upper subscapularis tear in Lafosse type 1 and type 2 with long head biceps tenotomy .
- group 2 (patient treated by arthroscopic repair with biceps tenotomy) (Active Comparator): repair of upper border subscapularis tear and doing biceps tenotomy
  Interventions: Procedure: skillful neglect Of upper subscapularis tear in Lafosse type 1 and type 2 with long head biceps tenotomy .; Procedure: arthroscopic repair Of upper subscapularis tear in Lafosse type 1 and type 2 with long head biceps tenotomy .

INTERVENTIONS:
Procedure: skillful neglect Of upper subscapularis tear in Lafosse type 1 and type 2 with long head biceps tenotomy . — The following technique will be utilized for confirm isolated or combined upper subscapularis border partial tear conservative treatment which is considered the standard technique.
  * Semisetting position under GA.
  * Standard shoulder arthroscopy with standard portals for RC repair.
  * Inspection of articular surface of rotator cuff and biceps tendon.
  * Bursectomy, visualization of all rotators.
  * Mobilization is done for associated rotator tears by shaver and radiofrequency device.
  * Both preoperative Statistics randomization that is used to determine which case will be repaired and intraoperative loss of tension of the elongated aspect of the tendon are used to confirm diagnosis and treatment of upper subscapularis border tear.
  * Skillful neglect to the tear.
  * Rotator repair technique by RC anchors
  * Biceps Tenotomy will be done in all cases by cutting of LHBT.
Procedure: arthroscopic repair Of upper subscapularis tear in Lafosse type 1 and type 2 with long head biceps tenotomy . — The following technique will be utilized for confirm isolated or combined upper subscapularis border partial tear repair which is considered the standard technique.
  * Semisetting position under GA.
  * Standard shoulder arthroscopy with standard portals for RC repair.
  * Inspection of articular surface of rotator cuff and biceps tendon.
  * Bursectomy, visualization of all rotators.
  * Mobilization is done for associated rotator tears by shaver and radiofrequency device.
  * Both preoperative Statistics randomization that is used to determine which case will be repaired and intraoperative loss of tension of the elongated aspect of the tendon are used to confirm diagnosis and treatment of upper subscapularis border tear.
  * Skillful neglect to the tear.
  * Rotator repair technique by RC anchors
  * Biceps Tenotomy will be done in all cases by cutting of LHBT.

SUMMARY:
The purpose of this study is to compare functional outcomes of Skillful Neglect & arthroscopic repair of upper border subscapularis tear in La fosse type 1 and type 2 with biceps tenotomy in non-athletes,30 shoulders subdivided randomly into 2 groups, 15 patients in group 1 (patient treated by skillful neglect with biceps tenotomy) and 15 patients in group 2 (patients treated by arthroscopic repair with biceps tenotomy)

DETAILED DESCRIPTION:
patients are randomized chosen then a shoulder arthroscope is done for all patients with biceps tenotomy but in group1 the investigators are neglecting the upper border tears and in group 2 the investigators are repairing upper border tears with anchors then after the procedure is completed the investigators will follow up by ASES score

ELIGIBILITY:
Inclusion Criteria:

* Patients with combined upper subscapularis border tear in Lafosse type 1 and type 2.

Exclusion Criteria:

* Glenohumeral arthritis.
* Patients with other intra-articular pathology like SLAP lesions.
* Neural damage (Brachial plexus injury).
* Revision cases.
* Patient with subscapularis border tear type 3, type 4, and type 5.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-09-26 (Estimated); Study Completion 2024-09-26 (Estimated)

PRIMARY OUTCOMES:
american shoulder elbow score | after 6months and 12 months
  scale that evaluates two dimensions of shoulder function: pain and performance in activities of daily living. Each of the two domains make up for 50 of the 100 points.

SECONDARY OUTCOMES:
Visual analogue score | Post operative 6months and 12 months
  subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

CONTACTS AND LOCATIONS:
Overall Officials: mohamed as abdallah, master, Principal Investigator — Ain Shams University; Amr Mo Abdelhady, Study Chair — Ain Shams University; Maged Mo Samy, Study Director — Ain Shams University; Mohamed Ha Sobhy, Study Director — Ain Shams University; Yahia Mo Haroun, Study Director — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No